CLINICAL TRIAL: NCT06969131
Title: The Current Role of Pentafecta Outcomes in Open and Laparoscopic Partial Nephrectomy for Localized Renal Tumors
Brief Title: Current Role of Pentafecta Outcomes in Open and Laparoscopic Partial Nephrectomy for Localized Renal Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Omar Ahmad Mohammed Bakheet, Assistant Lecturer of Urology, Faculty of Medicine, South Valley University, Egypt., South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVU/MED/URO016/2/22/5/400
Record Dates: First submitted 2025-04-27; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Pentafecta; Laparoscopic; Partial Nephrectomy; Renal Tumors
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Partial Nephrectomy (Experimental): Patients underwent open partial nephrectomy.
  Interventions: Procedure: Open Partial Nephrectomy
- Laparoscopic Partial Nephrectomy (Experimental): Patients underwent laparoscopic partial nephrectomy.
  Interventions: Procedure: Laparoscopic Partial Nephrectomy

INTERVENTIONS:
Procedure: Open Partial Nephrectomy — Patients underwent open partial nephrectomy.
  Arms: Open Partial Nephrectomy
Procedure: Laparoscopic Partial Nephrectomy — Patients underwent laparoscopic partial nephrectomy.
  Arms: Laparoscopic Partial Nephrectomy

SUMMARY:
This study aimed to identify predictive factors associated with the achievement of pentafecta outcomes following partial nephrectomy.

DETAILED DESCRIPTION:
Partial nephrectomy (PN) is widely considered the preferred treatment for clinical T1 (cT1) renal masses, primarily because it preserves kidney function more effectively than radical nephrectomy.

The trifecta metric includes three components: warm ischemia time (WIT) of ≤ 25 minutes or cold ischemia time (CIT) of ≤ 60 minutes, negative surgical margins, and the absence of perioperative major complications. The pentafecta expands upon these criteria by adding two additional parameters: preservation of ≥ 90% of the estimated glomerular filtration rate (eGFR) and no progression in chronic kidney disease (CKD) stage within 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* Patients who diagnosed with clinical T1 or T2a N0M0 renal tumors who were suitable candidates for partial nephrectomy

Exclusion Criteria:

* Severe and irreversible coagulopathy.
* Anatomically unfavorable tumor location.
* Extensive encasement of the renal pedicle.
* Diffuse invasion of the renal vein or central collecting system.
* Adjacent organ invasion consistent with stage cT4 disease.
* Regional lymphadenopathy (stage cTxN1), or anticipated retention of less than 20% of total nephron mass.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Predictor of pentafecta achievement | 12 months postoperatively
  Predictor of pentafecta achievement, such as smoking index, was recorded.

SECONDARY OUTCOMES:
Amount of blood loss | Intraoperatively
  Amount of blood loss was recorded.
Surgery duration | Intraoperatively
  Surgery duration was recorded.
Length of hospital stay | Till discharge from hospital (Up to one week).
  Length of hospital stay was recorded from admission till the discharge from hospital.
Intraoperative complications | Intraoperatively
  Intraoperative complications were recorded.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the visual analog scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable").
Analgesic requirements | 24 hours postoperatively
  Incidence of required analgesic was recorded.
Incidence of complications following surgery | 12 months postoperatively
  Incidence of complications following surgery were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley university, South Valley, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.